CLINICAL TRIAL: NCT07217899
Title: Phase II, Randomized, Double Blinded, Placebo Controlled Superiority Trial of Prophylactic Intravenous Calcium Gluconate to Decrease Blood Loss at Time of Cesarean Delivery in Pregnant Patients at High Risk for Uterine Atony
Brief Title: Prophylactic Intravenous Calcium Gluconate to Decrease Blood Loss at Time of Cesarean Delivery in Pregnant Patients at High Risk for Uterine Atony
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Molly Stout, Professor of Obstetrics and Gynecology Innovation, Associate Professor of Obstetrics and Gynecology and Section Head, Maternal Fetal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HUM00259931
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Blood Loss, Surgical; Blood Loss, Postoperative; Uterine Atony
Keywords: Cesarean delivery
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage; Uterine Inertia | interventions — Calcium Gluconate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This trial will include blinding of the subjects, investigators, and all direct care providers. There will be an anesthesiologist who is not involved in the clinical care of the patient who will be notified of the participant's randomization.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Randomized to receive intervention
  Interventions: Drug: Calcium Gluconate
- Arm 2 (Placebo Comparator): Randomized to receive placebo
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Calcium Gluconate — slow push intravenous administration of 2g calcium gluconate- 20 mL of 10% Calcium Gluconate in 55mL of IV fluid diluent, Normal Saline CaGluc concentration 26.7 mg/mL
  Arms: Arm 1
Other: Saline — slow push intravenous administration of 75 mL of IV
  Arms: Arm 2

SUMMARY:
This research study is being done to learn what effect a single dose of calcium gluconate will have on blood loss at the time of cesarean delivery in pregnancy patients at high risk for uterine atony.

DETAILED DESCRIPTION:
This study is FDA IND exempt

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Viable Intrauterine Pregnancy, Gestational Age ≥24 weeks
* Labor Converted to Cesarean Delivery at High Risk for Atonic Bleeding Defined as: Any exposure to oxytocin infusion for labor augmentation or induction prior to cesarean delivery
* Or Scheduled Cesarean Delivery at High Risk for Atonic Bleeding Defined as scheduled Cesarean-Section (CS) plus any one of:

  1. > 4 Prior deliveries
  2. General anesthesia
  3. Multifetal gestation
  4. Polyhydramnios diagnosed by ultrasound within 2 weeks
  5. Macrosomia ≥ 4000gms; estimated fetal weight by palpation or by ultrasound
  6. Fibroid uterus, defined as: Multiple ≥ 2cm intramural
  7. Any history of prior Primary postpartum hemorrhage (PPH)
  8. Platelets < 100,000 (but >50,000
  9. Placenta Previa
  10. Body Mass Index (BMI) ≥ 40

Exclusion Criteria:

* Non-English speaking
* Antenatal suspicion for placenta accreta spectrum
* History of allergic reaction to Calcium Gluconate
* Patients with hypertensive disorder of pregnancy receiving Magnesium Sulfate for seizure prophylaxis
* Underlying Renal Disease defined as Cr>1.0
* Known underlying cardiac condition
* Cardiac glycosides (Digoxin) within two weeks for maternal or fetal indication
* Treatment with a calcium channel blocker medication within 24 hours of screening
* Hypertensive disorder necessitating intravenous antihypertensive medication within 24 hours of screening
* Emergent case where study participation could impede care (judgement of obstetrician or anesthesiologist)
* Known hypercalcemia
* Concurrent use of any drugs that may cause hypercalcemia including

  1. Vitamin D
  2. Vitamin A
  3. Thiazide Diuretics
  4. Calcipotriene
  5. Teriparatide
* Ceftriaxone within 48 hours of screening
* Total Parenteral Nutrition (TPN) within 48 hours of screening
* Known Coagulopathy International Normalized Ratio (INR) ≥ 1.5
* Vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Quantitative Blood Loss (QBL) (continuous variable) administered at Delivery | Immediately following surgery
  Standardized volumetric assessment of blood loss during cesarean section

SECONDARY OUTCOMES:
Quantitative Blood Loss (QBL) (continuous variable) Total | 4 hours following surgery
  Standardized volumetric/gravimetric assessment of blood loss during cesarean section
Postpartum hemorrhage | 4 hours following surgery
  Quantitative blood loss ≥1000mL
Number of patients with a transfusion requirement | Calculated at 48 hours from delivery
  Any transfusion prior to discharge
Change in Hematocrit (HCT) | Preoperative day one, Postoperative day one
  Preoperative HCT and Post operative HCT measured though blood sample
Change in Hemoglobin (HGB) | Preoperative day one, Postoperative day one
  Preoperative HGB - Post operative HGB measured though blood sample
Number of participants with second line uterotonic requirements | Calculated at four hours from surgical end
  specific items of interest: Methylergonovine, Carboprost, or Misoprostol
Intensive Care Unit Admission | Within 48 hours of cesarean section
  Assessed using medical records
Additional hemostasis procedures | Within 48 hours of cesarean section
  Defined as requiring: Balloon Tamponade, Other atony device, B-Lynch, Uterine artery Ligation (Suture), Uterine Artery Embolization, Hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: AnneMarie Opipari, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No